CLINICAL TRIAL: NCT02191696
Title: Observational Study of ICD and Pacemaker Sensing in the Presence of IMED-4 Operation
Status: Completed | Type: Observational
Sponsor: Intersection Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-000050
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: IMED-4 recording

SUMMARY:
The purpose is to monitor far field sensing artifacts of CRM devices in the presence of the IMED-4

DETAILED DESCRIPTION:
The implanted CRM device will have shock therapy and rate sensor temporarily deactivated or placed in magnet mode during the time the IMED-4 is activated. The IMED-4 will be activated for a time not to exceed 15 minutes. During the time the IMED-4 is active, the CRM device programmer will print the voltage sensing of the implanted lead in real-time. The printout will be examined for the presence of far-field sensing artifacts.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with an active implantable CRM device
* Subjects > 18 years of age
* Subjects who are ambulatory not requiring assistance for ambulation
* Subjects who have been informed of the nature of the study and agree to its provisions and have provided written informed consent as approved by the IRB

Exclusion Criteria:

* Subjects who are pregnant or lactating or who have been pregnant within the past three months
* Subjects who have tattoos on the back in the electrode patch placement region
* Subjects who have had a past allergic reaction to adhesives
* Subjects who have poor general physical/mental health that, in the opinion of the investigator, will not allow the subject to be a good study candidate (i.e. other disease processes, mental capacity, substance abuse, shortened life expectance, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present for CRM device follow-up are possible candidates for the study and shall be screened for suitability based on the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
IMED-4 recordings | 6 months
  The primary endpoint is a collection of CRM device programmer printouts containing real-time lead sensing data from up to 40 unique subjects.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - North Coast Cardiology, Encinitas, California
  - Desert Heart, Palm Springs, California